CLINICAL TRIAL: NCT04920357
Title: CoVacc - Immune Response to Vaccination Against Covid-19, an Open Multicenter Phase IV Study
Brief Title: Immune Response to Vaccination Against Covid-19, a Follow up Study
Acronym: CoVacc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government); Värmland County Council, Sweden (Other Government); Örebro Läns Landsting (Other Government); Sormland County Council, Sweden (Other); Region Jämtland Härjedalen (Other)
Responsible Party: Sponsor
Other Study IDs: Eudra-CT2021-000683-30
Record Dates: First submitted 2021-05-31; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Vaccination; Infection; Covid19
Keywords: Immune response; Immunoglobulin G
MeSH Terms: conditions — Infections; COVID-19 | interventions — Vaccination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Periferal blood mononuclear cells (PBMC), plasma and sera.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID-19: Persons with a verified previous COVID-19 infection
  Interventions: Drug: Vaccination
- COVID-19 naive: Persons that have no history of COVID-19
  Interventions: Drug: Vaccination

INTERVENTIONS:
Drug: Vaccination — Persons that are vaccinated within the national and regional vaccine program are invited to participate in the follow-up study.

SUMMARY:
The study investigates the immune response after vaccination in individuals with and without pre-existing immunity to Coronavirus disease (COVID) -19. The participants are followed and sampled up to 4 years after vaccination. Blood samples are collected at different timepoints to analyze immune response.

The aim is to investigate the level of specific antibodies to Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) yearly, up to 4 years after vaccination.

DETAILED DESCRIPTION:
The main objective is to investigate if the antibody development to SARS-CoV-2 S protein differ after vaccination in those who have had a previous SARS-CoV-2 infection compared to Covid-19 naive individuals.

The secondary objective is to improve the understanding of the cellular and serological immune response after vaccination against COVID-19 in these groups.

Individuals with and without pre-existing immunity to COVID-19 are included in the study. They are included after informed consent at sites where they receive vaccines against COVID-19 within the national and regional vaccine campaign.

The study includes all approved COVID-19 vaccines with marketing authorization in Sweden.

Persons are enrolled after the first or second dose of vaccination and followed 4 years after vaccination. Blood is collected at inclusion and 3 months, 6 months, 1 year, 2 years, 3 years and 4 years after vaccination to assess the immune response.

Data on sex, age, body mass index, medical history and concomitant medication is collected.

The study is a follow-up study after vaccination and approved by the Swedish Medical Products Agency (EudraCT 2021-000683-30). Regular monitoring of the study is performed by the Clinical Trial unit at Umeå University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Consents to participate in the study
* Age ≥ 18 years

Exclusion Criteria:

* Age <18 years
* Incapable of giving informed consent
* Contraindication to vaccination
* Severe disease
* Ongoing treatment that is judged to affect the vaccine response (Does not include Rituximab which is allowed after individual consideration). Steroids > 15 mg orally per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with and without pre-existing immunity to Covid-19 that are vaccinated in the national and regional vaccine campaign.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in levels of specific IgG antibody against SARS-CoV-2 after vaccination over time. | 1 and 6 months, 1, 2, 3, and 4 years after vaccination.
  Levels of specific IgG antibody against SARS-CoV-2 will be measured as optical density, OD in a specific Spike-protein IgG ELISA at each time-point.
Change in proportion of participants with detectable specific IgG antibodies after vaccination over time. | 1 and 6 months, 1, 2, 3, and 4 years after vaccination
  Immune response will be measured as the proportion of participants (in % of all vaccinated individuals) with detectable specific IgG antibodies after vaccination at each time-point (in months after vaccination).

SECONDARY OUTCOMES:
Levels of markers for immune response after infection and vaccination against COVID-19 in COVID-naive versus COVID experienced individuals. | Change of markers for cellular and serological immune response over time measured at 1 and 6 months, 1, 2, 3, and 4 years after vaccination
  Levels of markers for cellular and serological immune response after COVID-19 vaccination e.g. specific antibodies, T- and B-cell memory.

CONTACTS AND LOCATIONS:
Overall Officials: Clas Ahlm, Prof, Principal Investigator — Umeå University
Locations (5):
- Sweden (5):
  - Mälarsjukhuset, Eskilstuna
  - Karlstad Central hospital, Karlstad
  - Örebro University hospital, Örebro
  - Östersund hospital, Östersund
  - Umeå University hospital, Umeå